CLINICAL TRIAL: NCT01790308
Title: Effect of Liraglutide Combined With Short-term CSII on Long-term Glycemic Remission and β Cell Function in Newly-diagnosed Type 2 Diabetic Patients
Brief Title: Effect of Liraglutide Combined With Short-term CSII on Long-term Glycemic Remission and β Cell Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, director of the endocrinology department of the First Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13450149260
Record Dates: First submitted 2013-02-06; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CSII (Active Comparator): continuous subcutaneous insulin infusion for 2-4 weeks
  Interventions: Drug: CSII
- Liraglutide (Active Comparator): continuous subcutaneous insulin infusion for 2-4 weeks combined with combined with Liraglutide 0.6mg/d for 2-4 weeks and 1.2mg/d for next 9 weeks
  Interventions: Drug: CSII; Drug: Liraglutide

INTERVENTIONS:
Drug: CSII — continuous subcutaneous insulin infusion for 2~4 weeks
Drug: Liraglutide — CSII for 2~4 weeks combined with Liraglutide 0.6mg/d for 1 month and 1.2mg/d for next 2 months
  Arms: Liraglutide

SUMMARY:
The purpose of this study is to investigate and evaluate the effects of liraglutide combined with short-term continuous subcutaneous insulin infusion(CSII) on long-term glycemic control and β-cell function in newly diagnosed type 2 diabetic patients.

DETAILED DESCRIPTION:
The purpose of this study is to investigate and evaluate the effects of liraglutide combined with short-term continuous subcutaneous insulin infusion(CSII)(1.CSII alone; 2.liraglutide combined with CSII) on long-term glycemic control and β-cell function in newly diagnosed type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed type 2 diabetes
* fasting blood glucose (FBG) level ranging from 7.0-16.7mmol/L
* body mass index (BMI) ranging from 21-35kg/m2
* antihypercaemic and antihyperlipidemic medication-naive patients

Exclusion Criteria:

* having any severe acute or chronic diabetic complications
* renal dysfunction, blood creatinine>150umol/L
* blood aminotransferase level rising up(more than 2 times of the upper normal limit of ALT)
* any severe cardiac disease including congestive cardiac failure, unstable angina or myocardial infarct in 12 months
* chronic or acute pancreatic disease
* severe systemic diseases or malignant tumor
* female patients incline to be pregnant
* being treated with corticosteriod, immunosuppressing drugs or cytotoxic drugs
* poor compliance

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
the percentage of the patients who maintain glucose control 1 year after short intensive therapy | 1 year

SECONDARY OUTCOMES:
the acute insulin response reflected β-cell function of different interventions in newly-diagnosed type 2 diabetic patients | 1 year
the remission rate differ from interventions in newly-diagnosed type 2 diabetic patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Li, MD, Principal Investigator — Ministry of Education